CLINICAL TRIAL: NCT03541382
Title: Community-led Distribution of HIV Self-tests: a Cluster Randomised Trial Investigating Uptake of HIV Testing and Linkage to Treatment and Prevention, Costs and Safety in Rural Malawi (HIV Self-Testing Africa [STAR])
Brief Title: A Cluster Randomised Trial of Community-led Distribution of HIV Self-tests in Rural Malawi (HIV Self-Testing Africa [STAR])
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Malawi-Liverpool-Wellcome Trust Clinical Research Programme (Other); Liverpool School of Tropical Medicine (Other); University College, London (Other); Population Services International (Other); UNITAID (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 14761
Record Dates: First submitted 2018-05-17; First posted 2018-05-30 (Actual); Last update posted 2020-08-11 (Actual); Status verified 2019-11

CONDITIONS: HIV/AIDS
Keywords: HIV; HIV Self-Testing; Malawi
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HIVST campaign arm (Active Comparator): Community representatives will be supported to plan and administer an HIVST campaign linked to HIV care and prevention services in their communities.
  Interventions: Device: OraQuick® HIV Self-Test
- SOC arm (No Intervention): Standard HTS will be provided by MoH at health facilities.

INTERVENTIONS:
Device: OraQuick® HIV Self-Test — Community leaders, including GVHs, Village Health Committee members, Village Development Committee members, and members of key community groups will participate in a workshop to facilitate planning of a HIVST campaign. Identified community distributors, who are unpaid volunteers from the community, will also receive a training package in HIVST promotion.
  Campaigns will be conducted over a short period (approximately seven days) and under a fixed budget. Community distributors will deliver HIVST kits free of charge to community members, and provide information on how to self-test and access the nearest clinic for linkage to confirmatory HTS, treatment and prevention. Distributors will also provide HIV prevention messages around serodiscordancy, treatment as prevention and VMMC.
  Arms: HIVST campaign arm

SUMMARY:
The aim of this study is to determine the benefits, costs and safety of community-led delivery of HIV self-testing (HIVST) kits in rural Malawi, with a focus on testing and linkage to care and prevention services among defined population sub-groups: men, adolescents aged 15-19 years old, and adults aged 40 years or older.

DETAILED DESCRIPTION:
RESEARCH QUESTION

Can community-led delivery of HIV self-tests be used to maximise public health and social benefits and reduce costs without introducing social harms?

RESEARCH AIMS AND OBJECTIVES

The broad aim is to determine the benefits, costs and safety of community-led delivery of HIVST kits in rural Malawi, with a focus on testing and linkage to care and prevention services among defined population sub-groups: men, adolescents aged 15-19 years old, and adults aged 40 years or older.

The specific objectives are to conduct a cluster randomised controlled trial to:

1. Establish the effectiveness of community-led HIVST campaigns on lifetime and recent HIV testing in predefined sub-groups.
2. Investigate the impact of community-led HIVST campaigns on: (a) population-level initiation of antiretroviral therapy (ART) and uptake of voluntary medical male circumcision (VMMC), (b) knowledge of HIV prevention, (c) stigma reduction
3. Explore how differences in community-led HIVST campaigns affect uptake of HIVST and linkage to care and prevention and values, attitudes and behaviours around HIVST.
4. Estimate the costs and cost-effectiveness of community-led HIVST campaigns compared to the standard of care (SOC).

RESEARCH DESIGN

The main study consists of a cluster-randomised trial evaluating the effectiveness of community-led HIVST campaigns on coverage of HIV testing and linkage to follow-on services compared to the Ministry of Health (MoH) SOC, facility-based HIV testing services (HTS). We are also interested in understanding the cost-effectiveness of community-led HIVST campaigns, and broader social benefits on stigma reduction.

The unit of randomisation is the Group Village Head (GVH), who are traditionally-appointed leaders that oversee a group of villages, and their catchments areas. Outcomes are measured through (i) household surveys in evaluation villages selected for each study cluster, and (ii) clinic records of patients coming from the study clusters.

For the primary outcome, measured using the households surveys, we assume that lifetime testing rates for adolescents aged 15-19 years old in the SOC arm are 35-50%, based on the recent Demographic and Health Survey. With 16 clusters per arm and 50 adolescents per cluster, we will have at least 90% power to detect a 20% absolute increase in lifetime testing using a coefficient of variation of outcomes (k) of 0.25. If k=0.3, for a 20% increase in lifetime testing, we would have 90% and 80% power with SOC testing rates of 35-40% and 45-55%, respectively. If the absolute increase in lifetime testing is lower at 15%, then for k=0.25 we would have 80% power for SOC testing rates of 35-40%. With adolescents making up 20-25% of the adult population, this will require 250 adults per cluster.

SUB-STUDIES

We will also be conducting a series of sub-studies related to the trial, including:

1. Process evaluation to monitor progress of the intervention and adherence to guidelines, and understand how differences in the context-driven intervention affect HIVST uptake and linkage to care and prevention.
2. Qualitative evaluation to explore which aspects of the community-led intervention were pivotal in affecting HIV testing and linkage outcomes and values, attitudes and behaviours around HIVST.
3. Economic evaluation to estimate costs, cost-effectiveness and cost-benefit per individual tested, newly diagnosed as HIV positive, started on ART and circumcised.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 15 years
* Residence in GVH catchment areas included in the intervention arm

Exclusion Criteria:

* Aged < 15 years old
* Not resident in GVH catchment areas included in the intervention arm

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 7880 (Actual)
Dates: Start 2018-10-08 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Percentage of self-reported lifetime testing in adolescents aged 15-19 years old | Measured 8-12 weeks post-intervention

SECONDARY OUTCOMES:
Percentage of self-reported testing in last 3 months in men aged ≥ 15 years | Measured 8-12 weeks post-intervention
Percentage of self-reported testing in last 3 months in adults aged ≥ 40 years | Measured 8-12 weeks post-intervention
Cumulative incidence of population-level ART uptake in adults aged ≥ 15 years over 6 months | Measured 6-months post-intervention
Measure of knowledge of HIV prevention methods | Measured 8-12 weeks post-intervention
Measure of HIV testing stigma. | Measured 8-12 weeks post-intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Malawi-Liverpool-Wellcome Trust Clinical Research Programme, Blantyre, Malawi

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Indravudh PP, Fielding K, Sande LA, Maheswaran H, Mphande S, Kumwenda MK, Chilongosi R, Nyirenda R, Johnson CC, Hatzold K, Corbett EL, Terris-Prestholt F. Pragmatic economic evaluation of community-led delivery of HIV self-testing in Malawi. BMJ Glob Health. 2021 Jul;6(Suppl 4):e004593. doi: 10.1136/bmjgh-2020-004593. PMID 34275869
- [Derived] Indravudh PP, Fielding K, Kumwenda MK, Nzawa R, Chilongosi R, Desmond N, Nyirenda R, Neuman M, Johnson CC, Baggaley R, Hatzold K, Terris-Prestholt F, Corbett EL. Effect of community-led delivery of HIV self-testing on HIV testing and antiretroviral therapy initiation in Malawi: A cluster-randomised trial. PLoS Med. 2021 May 11;18(5):e1003608. doi: 10.1371/journal.pmed.1003608. eCollection 2021 May. PMID 33974621
- [Derived] Indravudh PP, Fielding K, Kumwenda MK, Nzawa R, Chilongosi R, Desmond N, Nyirenda R, Johnson CC, Baggaley RC, Hatzold K, Terris-Prestholt F, Corbett EL. Community-led delivery of HIV self-testing to improve HIV testing, ART initiation and broader social outcomes in rural Malawi: study protocol for a cluster-randomised trial. BMC Infect Dis. 2019 Sep 18;19(1):814. doi: 10.1186/s12879-019-4430-4. PMID 31533646